CLINICAL TRIAL: NCT05756205
Title: A Randomized Controlled Low-intensity E-health Intervention by Midwives for Improving Mental Health in Pregnant Women
Brief Title: E-health Intervention for Improving Mental Health During Pregnancy Using Virtual Reality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/2018
Record Dates: First submitted 2023-02-08; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-11

CONDITIONS: Anxiety Depression; Pregnancy Related
Keywords: Pregnancy; Anxiety; Depression; Virtual Reality; Midwifery
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This will be a two-arm prospective, randomized, parallel-controlled clinical trial. 150 women will be recruited and screened during their pregnancy
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): The intervention will consist of an Immersive Virtual Reality (IVR) application with virtual reality goggles Oculus GO, to reduce anxiety during pregnancy. This application lasts 14 minutes by the use of mindfulness techniques based on breathing, mindfulness and passive muscle relaxation.
  Interventions: Device: Immersive Virtual Reality (IVR)
- Routine care (No Intervention): The control group will receive the usual follow-up pregnancy monitoring, without the e-health intervention.

INTERVENTIONS:
Device: Immersive Virtual Reality (IVR) — The intervention will consist of an Immersive Virtual Reality (IVR) application with virtual reality goggles Oculus GO, to reduce anxiety during pregnancy. This application lasts 14 minutes by the use of mindfulness techniques based on breathing, mindfulness and passive muscle relaxation. It consists of three modules that can be chosen completely or separately.
  The aspects that conform this intervention will be: information about, the most common perinatal mental health problems, exercises based on attention to breathing (mindfulness-relaxation), 6 weeks of duration, for 14 minutes a day, knowledge from involved personnel of the number of times the woman has connected and the time she has done the exercise, satisfaction questions to pregnant women after pregnancy, alerts to notify the principal investigator if there is a problem with e-health, and, finally, an email address to contact the principal investigator.
  Arms: Virtual Reality

SUMMARY:
Pregnancy-related anxiety and depression has received considerable attention worldwide. Mental health problems in pregnant women already since early weeks of gestation may have important consequences for the fetus. Current literature recommends the use of interventions based on new technologies for the treatment of mood disorders, already during the prenatal period. Adult pregnant women (weeks 12-14 of gestation) will be recruited and screened from different primary care centres in Catalonia, Spain. Women who pass the initial mental screening will be randomly allocated to the relaxation virtual reality intervention or control group. The intervention aims to improve mental state of pregnant women during pregnancy, work through breathing, mindfulness and muscle relaxation techniques.

DETAILED DESCRIPTION:
Background: Pregnancy-related anxiety and depression has received considerable attention worldwide. Mental health problems in pregnant women already since early weeks of gestation may have important consequences for the fetus. The necessity for more effective health care pathways, including some early interventions that reduce the overall burden of the childbearing situation, appears a key factor for a successful birth and care of the baby. The few studies focalized in interventions, are focused on delivery and post-partum, without taking into account the whole maternity process. Current literature recommends the use of interventions based on new technologies for the treatment of mood disorders, already during the prenatal period. There have been scarce well-designed intervention studies that test technological low-intensity interventions by midwives to address pregnant women's mental health, diminishing anxiety and depression during pregnancy.

Methods/design: Adult pregnant women (weeks 12-14 of gestation) will be recruited and screened from different primary care centres in Catalonia, Spain. Women who pass the initial mental screening will be randomly allocated to the relaxation virtual reality intervention or control group. The intervention aims to improve mental state of pregnant women during pregnancy, work through breathing, mindfulness and muscle relaxation techniques. Women in the control group will receive standard care offered by the public funded maternity services in Catalonia. The primary outcome measures will include the Edinburg Postnatal Depression (EPDS), State Trait Anxiety Inventory (STAI), Symptom Checklist-90 (SCL-90), and the Cambridge Worry Scale (CWS) instruments. Secondary outcome measures will include the Temperament and Character Inventory-Revised (TCI-R) and the Whooley and Generalized Anxiety Disorder-2 (GAD-2) questions. Routinely, pregnancy monitoring measures will also be evaluated.

Discussion: This study aims to test the efficacy of a low-intensity, midwife-led e-health intervention based on new technologies to work on women's anxiety and depression during pregnancy. The hypothesis is that that low-intensity mental health intervention during pregnancy, using an e-health (virtual reality) as a support tool, will be effective in reducing of anxiety, depressive symptoms, and improving satisfaction with pregnancy follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All women who control their pregnancy in the primary care centers of the Sexual and Reproductive Health Care (ASSIR; Atención a la Salut Sexual i Reproductiva) of Mutua Terrassa, Barcelona (Spain)
* The women must present a positive value in the mental health screening performed at the beginning of the pregnancy (weeks 12-14 of gestation).
* Verbal and written literacy understanding of Spanish
* ≥18 years old.

Exclusion Criteria:

* Women with diagnosed psychiatric pathology who are already being followed by the mental health team
* Women victims of gender-based violence who tested positive in the partner violence screen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Depression in pregnand women | 6 weeks
  Edingburg depression Scale (>9)
Anxiety in pregnand women | 6 weeks
  State trait anxiety inventory (>75%)

SECONDARY OUTCOMES:
Symptom checklist -90-R | 6 weeks
  Anxiety symptoms (>60%)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Jimenez Barragan, RN, RM, Principal Investigator — Fundació Assistencial Mutua Terrassa
Locations (2):
- Spain (2):
  - Fundació Assitencial Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitari Mútua Terrassa, Terrassa, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez-Barragan M, Del Pino Gutierrez A, Sauch Valmana G, Monistrol O, Monge Marcet C, Pallarols Badia M, Garrido I, Carmona Ruiz A, Porta Roda O, Esquinas C, Falguera Puig G. Immersive Virtual Reality eHealth Intervention to Reduce Anxiety and Depression in Pregnant Women: Randomized Controlled Trial. JMIR Hum Factors. 2025 Apr 30;12:e71708. doi: 10.2196/71708. PMID 40306641
- [Derived] Jimenez-Barragan M, Del Pino Gutierrez A, Garcia JC, Monistrol-Ruano O, Coll-Navarro E, Porta-Roda O, Falguera-Puig G. Study protocol for improving mental health during pregnancy: a randomized controlled low-intensity m-health intervention by midwives at primary care centers. BMC Nurs. 2023 Sep 7;22(1):309. doi: 10.1186/s12912-023-01440-4. PMID 37674184